CLINICAL TRIAL: NCT07107841
Title: Blinded, Randomized, Controlled, Trial to Evaluate the Efficacy and Safety of Autologous Hair Follicle Secretome for the Treatment of Androgenic Alopecia (Single Site)
Brief Title: Autologous Hair Follicle Secretome for Androgenic Alopecia (Single Site)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acorn Biolabs Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACN-401
Record Dates: First submitted 2025-07-31; First posted 2025-08-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Androgenic Alopecia; Alopecia; Baldness
Keywords: secretome; alopecia; Hair; stem cells; androgenic; androgenetic; Hormone; scalp; hair loss; baldness; bald; hair follicle; Acorn
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, double-blind
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-Secretome (Active Comparator): Intervention is autologous hair follicle-derived secretome diluted in saline
  Interventions: Other: Autologous Hair Follicle-Derived Secretome
- Placebo Control (Placebo Comparator): Placebo control is saline.
  Interventions: Other: Placebo Control

INTERVENTIONS:
Other: Autologous Hair Follicle-Derived Secretome — Hair follicles are plucked, cultured and the product is the resulting cell secretions (secretome) collected from the conditioned media.
  Other Names: aHFS
  Arms: Active-Secretome
Other: Placebo Control — The same saline used for diluting the active treatment in will be used as a control.
  Arms: Placebo Control

SUMMARY:
(SINGLE SITE Study) The purpose of this clinical trial is to evaluate the safety and efficacy of the use of an autologous hair follicle derived secretome for androgenous alopecia. The secretome will be injected into the scalp at baseline, and days 30, 90, 180, 270 and 365.

Hair growth will be quantitatively measured for density and thickness. PROs will also be collected from participants. This study will be run at a SINGLE SITE.

DETAILED DESCRIPTION:
(SINGLE SITE Study) Androgenic alopecia is a common condition causing hair loss and baldness in both men and women. Approximately 80 million men and women are affected by the condition in the US alone. Although there are a number of products on the market, both over the counter and prescribed, used for androgenic alopecia, they are only somewhat effective to slow the progression.

This trial will evaluate a new approach involving the injection of an autologous product made from the cellular secretions of hair follicles (secretome). Proteonomic analysis has demonstrated that this secretome contains anywhere from 2-22 times the bioactive components of platelet rich plasma (PRP) when compared within the same individual. The hypothesis is that repeat injections of autologous hair follicle-derived secretome will safely and effectively stimulate hair regrowth in men and women suffering from androgenic alopecia.

The trial is a double-blind, randomized, placebo controlled study in 60 patients who are on a stable (>6 months) regimen of minoxidil and 5 alfa-reductase inhibitors. The injections will be delivered at baseline (day 0), 30, 90, 180, 270 and 365 days as follows:

* Each vial of secretome will be diluted with 2ml of saline
* Each quadrant of the affected scalp will receive one vial of secretome
* Injections will be delivered in a grid-like pattern with injections spaced ~1cm apart
* Approximately 20 injections (0.1ml/injection) will be delivered to each alopecia affected quadrant

ELIGIBILITY:
Inclusion Criteria

* SUBJECTS MUST BE ON A STABLE COURSE OF MINOXIDIL (ORAL OR TOPICAL) AND/OR 5-ALPHA REDUCTASE INHIBITORS. THEY MUST HAVE BEEN ON THE SAME 5-ALPHA REDUCTASE INHIBITOR FOR ≥12 MONTHS PRIOR TO BASELINE.
* FEMALE SUBJECTS MUST NOT BE ON HAIR GROWTH MEDICATIONS OR TOPICALS FOR ≥6 MONTHS PRIOR TO BASELINE.
* TESTOSTERONE REPLACEMENT THERAPY (TRT) IN ANY FORM (E.G. DEPO-, INJECTABLE, TOPICAL, PATCHES, NASAL GEL, ORAL, PELLET ETC.) IS ALLOWED AS LONG AS SUBJECT HAS BEEN ON A STABLE COURSE (IN THE OPINION OF THE INVESTIGATOR) OF TRT FOR ≥12 MONTHS.
* Biological sex: Male and Female (up to n=20 males and up to n=10 females will be in each arm for a total of up to n=40 males and up to n=20 females)
* Age: ≥18 - 65 years
* Subjects with Androgenic alopecia
* No intention to start new hair growth medications and no intention to change the dosage or usage of minoxidil or 5-alpha reductase inhibitors until the end of their participation in the trial.
* Competent and willing to provide written, informed consent to participate in all study activities.
* Willing and able to tolerate multiple injections of the study product.
* Must be able to attend all study related clinical visits.
* Willing to maintain the same hair style as at the Screening Visit for the duration of the study.
* Must be willing to have small (diameter similar to a pencil lead) UV (invisible) or red colored tattoo dots applied to scalp (up to 5) and touch up tattoos if necessary. UV tattoo dots only show under black light. Subjects will chose UV or red.

Exclusion Criteria

* Subjects with clinical diagnosis of alopecia areata or other non-androgenic forms of alopecia.
* Active skin disease (Psoriasis or severe seborrheic dermatitis) of the scalp
* Scalp infection
* Severe active systemic infection
* Cuts or abrasions on the scalp
* History of surgical hair restoration in the last 12 months.
* Current or recent (within last 5 years) malignancy (except basal cell and squamous cell skin cancers)
* History of systemic chemotherapy or radiation
* History of thyroid dysfunction
* History of autoimmune disorder (specifically Graves disease, Hashimoto thyroiditis, or systemic lupus erythematosus)
* Continuous/daily use of nonsteroidal anti-inflammatory or Vitamin E, unless discontinued within 7 days before 1st treatment and only used as needed through the trial period.
* Use of any medications that potentially cause drug-induced hair loss (e.g., depo-testosterone, haloperidol, methotrexate, methylprednisolone, prednisone, testosterone, divalproex sodium) within the last 3 months.
* Known allergy or sensitivity to tattoo ink.
* Current anticoagulant therapy (heparins; factor Xa inhibitors; direct agents such dabigatran, rivaroxaban, apixaban, edoxaban and betrixaban; warfarin/coumarins)
* Significant tendency to develop keloids or hypertrophic scarring
* Subjects unable to communicate with the investigator and staff
* Any health condition that in the investigator's opinion should preclude participation in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Target Area Hair Counts (TAHC) | 180 Days after Baseline
  Non-vellus TAHC is the number of non-vellus (terminal) hairs within 1 cm² scalp
Safety | 180 days from Baseline
  Incidence rates of treatment-related adverse events compared between the active and placebo arm

SECONDARY OUTCOMES:
Mean Total Hair Density (vellus and non-vellus/terminal) | 30, 90, 270 and 365 days
  Mean Total Hair Density (vellus and non-vellus/terminal): measured by Trichoscan device
Patient Satisfaction | 30, 90, 270 and 365 days
  Patient satisfaction collected using a 5 point Likert scale
Hair thickness improvement | 30, 90, 180, 270 and 365 days
  Hair thickness improvement measured by Trichoscan device
Patient Global Impression of Change (PGIC) | 180 and 365 days
  Patient rated improvement in alopecia based on comparison of Baseline to follow-up time point

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Campbell, PhD, Study Director — Acorn Biolabs
Locations (1):
- Ziering Medical, West Hollywood, California, United States

IPD SHARING:
Plan to Share IPD: No
This is a proof of concept study on a unique product unlike others so there is no reason to share IPD